CLINICAL TRIAL: NCT05022810
Title: A Randomized, Open Label, Single Center, Single Dose, Two Period, Two Sequence, Crossover Bioequivalence Study of Paracetamol in a New Pediatric Paracetamol Oral Suspension Compared to a Marketed Paracetamol Oral Suspension (Panadol Baby & Infant) in Healthy Adult Subjects
Brief Title: A Bioequivalence Study of a New Paracetamol Oral Suspension 24mg/ml Compared to the Marketed Paracetamol Oral Suspension (Panadol Baby and Infant 24mg/ml) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 215262; 2021-000900-40 (EudraCT Number)
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: This is a 2-arm, single center, single dose, open-label, randomized, two sequence, two-period crossover, bioequivalence study in healthy adult subjects, separated by one wash-out period of at least 72 hours.
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): Participants will receive a single oral dose of either New Paracetamol Oral Suspension (24 mg/ml) or Panadol B&I Oral Suspension (24 mg/ml paracetamol) on Day 1 (Period 1) and Day 4 (Period 2) under fasting conditions as per the randomization schedule. A wash out period of at least 72-hour will be maintained between each treatment period.
  Interventions: Drug: New Paracetamol Oral Suspension (24 mg/ml)
- Reference Drug (Active Comparator): Participants will receive a single oral dose of either New Paracetamol Oral Suspension (24 mg/ml) or Panadol B&I Oral Suspension (24 mg/ml paracetamol) on Day 1 (Period 1) and Day 4 (Period 2) under fasting conditions as per the randomization schedule. A wash out period of at least 72-hour will be maintained between each treatment period
  Interventions: Drug: Panadol B&I Oral Suspension (24 mg/ml paracetamol)

INTERVENTIONS:
Drug: New Paracetamol Oral Suspension (24 mg/ml) — After an overnight fasting for at least 10 hours, New Paracetamol Oral Suspension (24 mg/ml) in a volume of 42 ml will be administered orally via a single use syringe by a trained study person to the study participants as per the randomization schedule in each period.
  Arms: Test Drug
Drug: Panadol B&I Oral Suspension (24 mg/ml paracetamol) — After an overnight fasting for at least 10 hours, Panadol B&I Oral Suspension (24 mg/ml paracetamol) in a volume of 42 ml will be administered orally via a single use syringe by a trained study person to the study participants as per the randomization schedule in each period.
  Arms: Reference Drug

SUMMARY:
The objective of the study is to compare the bioequivalence of a New Paracetamol Oral Suspension 24 milligram/milliliter (mg/ml) with that of an already approved Paracetamol (24 mg/ml) Oral Suspension (Panadol Baby & Infant) when administered to healthy volunteers under fasting condition. Pharmacokinetic parameters will be calculated from plasma concentration data. The rate and extent of absorption of the formulations will be compared.

DETAILED DESCRIPTION:
This will be a 2-arm, single center, single dose, open-label, randomized, two-sequence, two period crossover, bioequivalence study in healthy adult participants. Participants will be screened for eligibility within 15 days prior to dosing. Participants will receive each of the two study treatments in fasted state during a 6-day (5-overnight stay) residential period at the study site. Participants will receive both treatment regimens in a randomized order with a 72-hour washout period between each dose. During each treatment period, a total of 21 blood samples will be collected which will include a pre-dose blood sample 1 hour before dosing and 20 post-dose blood samples at 5, 10, 20, 30, 40, 50, 60, 80, 90, 120, 150, 180 minutes, 4, 5, 6, 8, 10, 12, 14, 16 hours, for bioanalytical analyses of paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan, laboratory tests, study restrictions and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, as determined by medical evaluation, including medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* A participant with a Body Mass Index (BMI) of 18.5 to 30.0 kg/m^2; and a total body weight >50 kg
* Female participants of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for 7 days after the last dose of assigned treatment.
* Participant with two consecutive negative tests for active COVID-19, separated by > 24 hours.
* Czech citizenship

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSKCH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days before dosing.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is pregnant as confirmed by a positive hCG laboratory test or intending to become pregnant over the duration of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients. This includes paracetamol and excipients in the products e.g. sorbitol, maltitol glycerol etc.
* A participant unwilling or unable to comply with Lifestyle Considerations.
* Diagnosis of long QT syndrome or QTc > 450 msec for males and > 470 msec for females at screening.
* A participant with evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance but not limited to any of the following:
* History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling or gastric banding (note: this is not applicable for minor abdominal surgery without significant tissue resection, e.g., appendectomy and herniorrhaphy)
* History of inflammatory bowel disease
* History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine (≥ 123 μmol/l) or urea (≥ 8.9 mmol/L) or the presence of clinically significant abnormal urinary constituents (e.g. albuminuria);
* History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A candidate will be excluded if more than one of the following lab value deviations are found: 1) AST/SGOT (≥ 1.2 ULN), ALT/SGPT (≥ 1.2 ULN), 2) GGT (≥ 1.2 ULN), ALP (≥ 1.2 ULN), 3) bilirubin (≥ 1.2 ULN) or CK (≥ 3 ULN). A single deviation from the above values is acceptable and will not exclude the candidate, unless specifically advised by the Investigator;
* Evidence of urinary obstruction or difficulty in voiding at screening.
* History or clinical evidence at screening of pancreatic injury or pancreatitis
* A participant with history of regular alcohol consumption exceeding 18 g (women) or 35 g (men) of pure alcohol per day, i.e. 1 drink/day for women or 2 drinks/day for men (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening
* Participant reported regular consumption of > 5 cups of coffee or tea per day (or equivalent consumption of ≥ 500 mg xanthine per day using other products)
* Positive results in any of the virology tests for HIV-Ab, HCV-Ab, HBsAg and HBc-Ab (IgG + IgM)
* Allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the Investigator's opinion may pose a risk to the candidate.
* Any condition not identified in the protocol that in the opinion of the Investigator would confound the evaluation and interpretation of the study data or may put the participant at risk
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study
* Use of any medication (including over-the-counter medications, vitamins, herbal remedies, dietary supplements) within 2 weeks prior to admission to the unit or within less than 10 times the elimination half-life of the respective drug (whichever is longer) or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:
* systemic contraceptives and hormone replacement therapy, as long as female participant is on stable treatment for at least 3 months and continues treatment throughout the study;
* occasional use of ibuprofen 200 mg (up to 1200 mg daily) or equivalent analgesic
* Participant reports consumption of any drug metabolizing enzyme (e.g. CYP3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (e.g. broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort etc.) within 2 weeks prior to admission to the unit
* Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 90-140 mmHg for systolic BP and/or 60-90 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
* Body temperature is consistently out of the range of 35.4-37.3°C at screening, at check-in or during the study.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within 2 weeks prior to screening till admission to the unit
* A participant with a positive urine drug screen, alcohol breath test at screening and on day of admission to the unit
* Smokers, defined as the use of tobacco products during the 3 months prior to screening till admission to the unit or a positive urine cotinine test at screening
* Performance of strenuous physical exercise (body building, high performance sports) from 2 weeks prior to admission to the unit
* Donation or loss of at least 500 mL of blood within 90 days or any donation of plasma or platelets from 2 weeks prior to admission to the unit
* Getting a tattoo, body piercing or any cosmetic treatment involving skin penetration within 90 days before the screening till admission to the unit, unless evaluated by Investigator as non-significant for inclusion in the study
* Participant with signs and symptoms suggestive of COVID-19 (i.e. fever, cough, etc.) from 2 weeks prior to screening till admission to the unit
* Participant with known COVID-19 positive contacts in the past from 2 weeks prior to screening till admission to the unit
* Participants who were hospitalized for COVID-19 related reasons

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in Czech Republic.
Pre-assignment Details: A total of 61 participants were enrolled into the study, of which 21 were screen failures, 5 were not assigned to any treatment and 35 were randomized to the study treatment. All the randomized participants completed the study.
Groups:
- Test Drug/Reference Drug: Participants received new paracetamol suspension (Test drug) orally as a single 42 milliliter (mL) (1 gram [g] paracetamol) dose in treatment period 1. In treatment period 2, participants received marketed paracetamol suspension (Reference drug) orally as a single 42 mL (1 g paracetamol) dose. There was a washout period of 3 days between two treatment periods.
- Reference Drug/Test Drug: Participants received marketed paracetamol suspension (Reference drug) orally as a single 42 mL (1 g paracetamol) dose in treatment period 1. In treatment period 2, participants received new paracetamol suspension (Test drug) orally as a single 42 mL (1 g paracetamol) dose. There was a washout period of 3 days between two treatment periods.
Period: Period 1 (2 Days)
Arm/Group | Test Drug/Reference Drug | Reference Drug/Test Drug
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Washout Period (3 Days)
Arm/Group | Test Drug/Reference Drug | Reference Drug/Test Drug
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Period 2 (2 Days)
Arm/Group | Test Drug/Reference Drug | Reference Drug/Test Drug
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population - Comprised of all randomized participants who received at least one study medication.
Groups:
- Test Drug/Reference Drug: Participants received new paracetamol suspension (Test drug) orally as a single 42 mL (1 g paracetamol) dose in treatment period 1. In treatment period 2, participants received marketed paracetamol suspension (Reference drug) orally as a single 42 mL (1 g paracetamol) dose. There was a washout period of 3 days between two treatment periods.
- Total: Total of all reporting groups
Arm/Group | Test Drug/Reference Drug | Reference Drug/Test Drug | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.7 (6.7) | 30.6 (7.8) | 30.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 12 | 8 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Plasma Concentration [AUC] Versus Time Curve Calculated From Time Zero to the Last Measurable Sampling Time Point (Tlast) (AUC [0-tlast])
Description: Blood samples were collected at the indicated time points for the analysis of AUC (0-tlast). Pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (-1 hour) and 0.08, 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.33, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 14, 16 hours Post dose.
Population: PK Population - Comprised of participants in the 'Safety' population who complete the two periods and who have no major protocol deviations concerning PK.
Measure: Mean (Standard Deviation); unit: microgram*hour/mL
Groups:
- Test Drug: Participants received new paracetamol suspension (Test drug) orally as a single 42 mL (1 g paracetamol) dose in treatment period 1 and in treatment period 2.
- Reference Drug: Participants received marketed paracetamol suspension (Reference drug) orally as a single 42 mL (1 g paracetamol) dose in treatment period 1 and in treatment period 2.
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 35 | 35
microgram*hour/mL | 47.18 (9.3702) | 48.12 (10.749)

2. Primary Outcome: The Time of the Maximum Observed Post-dose Concentration (Tmax)
Description: Blood samples were collected at the indicated time points for for the analysis of tmax. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Median (Full Range); unit: hour
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 35 | 35
hour | 1 [0.33 to 4.00] | 1 [0.50 to 2.00]

3. Primary Outcome: The Maximum Observed Post-dose Concentration (Cmax)
Description: Blood samples were collected at the indicated time points for for the analysis of Cmax. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: microgram/mL
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 35 | 35
microgram/mL | 11.63 (2.2598) | 11.59 (2.4865)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Calculated From Time Zero to Infinity [AUC (0-inf)]
Description: AUC (0-inf) = AUC (0-tlast) + Clast/ λz, where Clast is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples were collected at the indicated time points for for the analysis of AUC (0-inf). PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: microgram*hour/mL
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 35 | 35
microgram*hour/mL | 49.14 (9.6926) | 50.18 (11.312)

5. Secondary Outcome: Percentage of AUC (0-inf) Obtained by Extrapolation (%AUCex)
Description: %AUCex = (1- [AUC0-tlast/AUC0-inf]*100). Blood samples were collected at the indicated time points for for the analysis of %AUCex. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Percentage of AUC
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 35 | 35
Percentage of AUC | 3.981 (1.5695) | 4.056 (1.5082)

6. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: λz is computed as the slope of the regression line of ln (concentration) verses time. Blood samples were collected at the indicated time points for for the analysis of λz. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 35 | 35
1/hour | 0.2061 (0.06784) | 0.2059 (0.06396)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from screening up to Day 7.
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout product, whether or not considered related to the study product.
Arm/Group | Test Drug | Reference Drug
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT05022810/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT05022810/SAP_001.pdf